CLINICAL TRIAL: NCT07096102
Title: Efficacy of a Health Empowerment Theory Based Health Information Literacy Promotion Intervention in Individuals With Metabolic Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meihua Ji (Other)
Collaborators: The Luhe Teaching Hospital of the Capital Medical University (Other)
Responsible Party: Sponsor-Investigator, Meihua Ji, Associate Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Main_RCT_ENRICH
Record Dates: First submitted 2025-07-16; First posted 2025-07-31 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Metabolic Syndrome (MetS)
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENRICH Intervention Group (Experimental): A 6-week intervention programme was implemented for the health information literacy enhancement group, once a week, with each intervention lasting 30-40min, to enable the study participants to actively practice healthy behaviours through intervention techniques such as health awareness awakening, social resource building, and health-related skill empowerment, in order to enhance the health information literacy of the study participants, and ultimately to enable the study participants to perceive health in a programmatic manner.
  Interventions: Behavioral: ENRICH Group
- Routine Care Group (Active Comparator): Receiving routine health education: distributing health education handbooks on metabolic syndrome and metabolic diseases, establishing WeChat groups, and delivering regular weekly health knowledge.
  Interventions: Behavioral: Routine Care Group

INTERVENTIONS:
Behavioral: ENRICH Group — Participants will undertake a six-week programme to enhance their health information literacy. The specific details are as follows: (1) Capacity Building on Health Information Management via Health Education Based on the Health Empowerment Theory:①Strengthening skills related to Health Information Literacy; ②Training on Medication Management Skills;③ Practice of Self-Monitoring Skills;④Education on Diet and Exercise Management Knowledge. (2) Health Behavior Motivation Management Based on the Health Empowerment Theory:① Personalized Goal Setting;②Behavioral Incentives and Feedback;③Construction of Peer Support Networks;④Demonstration Effect of Role Models. (3) Health Management Support System Based on the Health Empowerment Theory:①Online Dynamic Monitoring;②Family-Community Collaborative Support;③Digital Monitoring Platform;④Continuous Supply of Resources.
  Arms: ENRICH Intervention Group
Behavioral: Routine Care Group — ①Distribute 3-5 push publics on screening health information and health disinformation in the first week；②Distribute 3-5 push publics on medicine knowledge in the second week；③Distribute 3-5 push publics on self-monitoring knowledge in the third week；④Distribute 3-5 publics on exercise knowledge in week 4；⑤Distribute 3-5 push publics on dietary knowledge in week 5 and week 6.
  Arms: Routine Care Group

SUMMARY:
The ENRICH study is aimed to Enpower patieNts with metabolic syndrome (Mets) to increase their Risk perception and to acquire health Information necessary for Capability building and promotion of Health information literacy, as well as health outcomes. The purpose of this clinical trial is to evaluate the efficacy of this health information literacy promotion intervention based on Health Empowerment Theory in individuals with metabolic syndrome. The study aims to answer the following questions:

Does the intervention improve health information literacy among study participants? Does the intervention lead to better health outcomes, including weight, waist circumference, BMI control, and metabolic health indicators (blood pressure, blood glucose, glycated hemoglobin, and blood lipids)?

Participants will:

Undergo the intervention program for 6 weeks (face to face and online) and will be assessed regularly to monitor changes in terms of their level of health information literacy and health outcomes.

DETAILED DESCRIPTION:
Participants enrolled in the ENRICH study is planned to receive activities related to:

1. Health information management ability education based on health empowerment theory:①health information literacy intensive training;②medication management skills training;③self-monitoring skills practice;④diet and exercise management knowledge education.
2. Health behaviour motivation management based on health empowerment theory:①personalized goal setting: set learning goals with patients and clarify the weekly health information literacy improvement plan;②behavioural incentives and feedback: give spiritual recognition and physical rewards to patients who complete the health punch card on time and meet the monitoring targets;③peer support network construction: set up a discussion group to encourage patients to share their experiences in diet management and exercise practice, and enhance their knowledge of diet and exercise through group interaction;④Role model demonstration effect: patients with high health information literacy and remarkable self-management effects are set up as role models, and are invited to share their success stories.
3. Health management support system building based on the theory of health empowerment: ①online dynamic supervision: weekly Q&A sessions through WeChat groups to address issues such as health information screening, medication use, and interpretation of monitoring data;② collaborative family-community support: inviting family members to join the health management group to assist in dietary planning, supervise the implementation of exercise, and linking with the community health service centres to provide personalized guidance;③digital monitoring platforms Digital monitoring platform: Using the Concordia Medical Weight Loss applet and diet management WeChat group to push customised health advice;④Continuous supply of resources: Regularly updating links to authoritative channels, such as the website of the State Drug Administration and the China Public Health Network, to ensure that patients have access to reliable health information.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and ≤ 75 years old;；
* Patients diagnosed with metabolic syndrome (meeting ≥3 criteria):
* Waist circumference ≥ 90 cm (men) / ≥ 85 cm (women)
* Fasting glucose ≥ 6.1 mmol/L or OGTT 2h-glucose ≥ 7.8 mmol/L and/or diabetes treatment
* Blood pressure ≥ 130/85 mmHg and/or hypertension treatment
* Fasting triglycerides (TG) ≥ 1.70 mmol/L
* Fasting HDL-C < 1.04 mmol/L；
* Aware of the condition, have basic reading and language communication skills, and voluntarily participate in this study

Exclusion Criteria:

* Patients with severe liver and kidney dysfunction, cancer, severe cardiovascular and cerebrovascular diseases, gout, etc., which seriously endanger life, have abnormal nutritional status and require special diet;
* Pregnant patients；
* Patients with a history of mental illness and cognitive impairment；
* Those currently participating in other research projects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-08-31 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Health Information Literacy | Measurements will be conducted before the intervention (baseline measurement), at the end of the intervention (immediate measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  Health information literacy (HIL) is essential to assist individuals in health decision-making. In this study, health information literacy will be measured using the Health Information Literacy Self-rating Scale.A 5-point Likert scale was used, with scores ranging from 1-5 for 'strongly disagree to 'strongly agree', and a total scale score ranging from 0-29, with higher scores indicating higher levels of health information literacy. In the original study, the Cronbach's a coefficient for HILSS was 0.847, and the Cronbach's a coefficients for the dimensions was 0.783～0.917.
Chronic Patient Self-Management Questionnaire | Measurements will be conducted before the intervention (baseline measurement), at the end of the intervention (immediate measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  The Self-Management Questionnaire for Chronic Patients used to assess the self-management level of patients with chronic diseases. The scale includes five aspects: dietary habits, exercise management, medication adherence, emotional management, and family and social support, and adopts the Likert 5-point rating method. The questionnaire consists of 20 multiple choice questions with a total score of 100 points. The scoring criteria are: between 20 and 60 points is a poor level of self-management; between 60 and 80 points is a medium level of management; between 80 and 100 points is a high level of self-management. The Cronbach's a coefficient of the scale is 0.957.
Glycosylated Hemoglobin（HbA1c ) | Measurements will be conducted before the intervention (baseline measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  The glycosylated hemoglobin level is determined by past, rather than immediate, blood glucose concentrations. The glycosylated hemoglobin concentration is generally considered to be a valid reflection of the average blood glucose level over the past 8 to 12 weeks.
Total Cholesterol（TC）, Triglyceride（TG）, High Density Lipoprotein-Cholesterol（HDL-C）, Low-Density Lipoprotein Cholesterol（LDL-C） | Measurements will be conducted before the intervention (baseline measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  1. Total cholesterol is the sum of the cholesterol in all lipoproteins in the blood. If this indicator is high, it may be related to physiological factors such as smoking and stress, or disease factors such as familial hypercholesterolaemia and diabetes mellitus.
  2. Triglyceride (TG) is a type of fat in the blood, which is mainly derived from fat in food and synthesised by the liver. High levels of triglycerides are one of the risk factors for cardiovascular disease.
  3. High-density lipoprotein cholesterol (HDL-C) is a beneficial cholesterol that removes LDL cholesterol from the blood vessels and reduces the risk of cardiovascular disease.
  4. Low-density lipoprotein cholesterol (LDL-C) is a harmful cholesterol and is one of the major risk factors for cardiovascular disease.The higher the LDL cholesterol level, the greater the risk of cardiovascular disease.
General Physical Examination- Height | Measurements will be conducted before the intervention (baseline measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  The participants shall be measured bareheaded and barefoot using a vertical stadiometer with an accuracy of 0.1 cm. During the measurement process, each indicator is required to be measured using uniform standards and instruments.
General Physical Examination- Weight | Measurements will be conducted before the intervention (baseline measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  The measurement shall be conducted using a metrologically certified weighing scale, with the participant standing calmly at the center of the platform, distributing weight evenly on both legs, and measured bareheaded and barefoot. During the measurement process, each indicator is required to be measured using uniform standards and instruments.
General Physical Examination- Body Mass Index（BMI） | Measurements will be conducted before the intervention (baseline measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  According to the internationally recognized BMI calculation formula:
  BMI = weight (kg) / height (m)²
General Physical Examination- Waist Circumstance | Measurements will be conducted before the intervention (baseline measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  The measurement shall be performed by marking the midpoint between the lower edge of the rib cage at the midaxillary line and the iliac crest on both sides. A flexible measuring tape shall be placed horizontally around the body at the marked points, maintaining gentle contact with the skin without compression. The reading shall be taken at the end of normal expiration. During the measurement process, each indicator is required to be measured using uniform standards and instruments.
General Physical Examination- Blood Pressure | Measurements will be conducted before the intervention (baseline measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  Blood pressure measurement shall be performed after the subject has rested quietly in a seated position for at least 5 minutes, with the upper arm positioned at heart level. Using a standard sphygmomanometer, two consecutive measurements of upper arm blood pressure shall be taken at 1-2 minute intervals, with the final result recorded as the average of the two readings. During the measurement process, each indicator is required to be measured using uniform standards and instruments.
General Physical Examination- Blood Glucose | Measurements will be conducted before the intervention (baseline measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  The subject's meal consumption status and timing shall be inquired and recorded, followed by random fingertip blood glucose measurement using a standardized glucometer. During the measurement process, each indicator is required to be measured using uniform standards and instruments.

SECONDARY OUTCOMES:
Health Literacy | Measurements will be conducted before the intervention (baseline measurement), at the end of the intervention (immediate measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  Health literacy refers to an individual's ability to obtain, process, and understand basic health information and services, and to make appropriate health decisions. Compared with health information literacy, the concept and scope of health literacy are more general and broader.In this study, the Newest Vital Sign scale will be used to assess individuals' overall health literacy levels. The measure has six questions assessing a person's reading, numeracy, and comprehension based on an ice cream nutritional label. 1 point for each correct answer, 6 questions in total, total score 0-6 points, the higher the score the higher the health literacy. The internal consistency (Cronbach's a) was 0.76.
Health Problem Solving | Measurements will be conducted before the intervention (baseline measurement), at the end of the intervention (immediate measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  The Chinese version of the Health Problem-Solving Scale consists of 6 dimensions: rational/effective problem-solving, positive positive transfer problem-solving, avoidance problem-solving, impulsive/careless problem-solving, negative transfer/learning, and negative motivation/attitude. It includes 30 items. The Likert 5-point scoring method was used, with the lowest score being 0 and the highest score being 4. The higher the score, the better the health problem solving ability. The content validity index of the scale is 0.970, the content validity index of the items ranges from 0.830 to 1.000, the Cronbach's a coefficient is 0.911, and the Cronbach's a coefficients of each dimension range from 0.715 to 0.839.
Chronic Illness Resources | Measurements will be conducted before the intervention (baseline measurement), at the end of the intervention (immediate measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  The Chronic Illness Resource Survey (CIRS) consists of 19 items measuring six aspects of social resources: individuals, family and friends, healthcare team, community, media policy and community organisations. The scale is scored on a 5-point Likert scale, ranging from 1 to 5. Higher scores indicate greater access to or use of resources. The scale had good reliability in the original study, with a Cronbach's a coefficient of 0.820, and an overall Cronbachs a coefficient of 0.845 in the Chinese population.
Chronic Disease Self-Efficacy Scale | Measurements will be conducted before the intervention (baseline measurement), at the end of the intervention (immediate measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  The scale consists of 6 items in 2 dimensions, including patients' symptom management self-efficacy (measured by items 1-4) and patients' disease co-management self-efficacy (measured by items 5-6). The scale was rated on a 10-point positive scale, with a minimum score of 1 indicating that the patient was not at all confident in health self-management, a maximum score of 10 indicating that the patient was confident in health self-management, and a total score of the average of the 6 entries. The higher the score, the better. The original version of the scale had a Cronbach's a coefficient of 0.91.
Knowledge of Metabolic Syndrome Scale (K-MS scale) | Measurements will be conducted before the intervention (baseline measurement), at the end of the intervention (immediate measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  The scale consists of 10 entries in 3 dimensions: disease definition, hazards, and prevention and treatment (all single-choice questions with 5 choices each). The scale is scored by calculating the percentage of correct answers, with one correct answer counting for 10 points and a total score of 0-100, with higher scores being better. The total Cronbach's a coefficient of the scale was 0.69, the Cronbach's a coefficient of each entry was 0.63-0.73, the re-test reliability was 0.56 (P=0.0002), the content validity (CVI) was 98.1%, and the measurements were in line with the hypothesised construct validity (P<0.0001).
Nutrition Literacy | Measurements will be conducted before the intervention (baseline measurement), at the end of the intervention (immediate measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  The Food and Nutrition Literacy Questionnaire, developed by the School of Public Health at Peking University, will be used for assessment. The current status of nutrition literacy includes four dimensions: knowledge and concepts related to food, selecting food, preparing food, and consuming food. The questionnaire has a score of 100 points, and the critical value of this questionnaire is 80 points, and a score of 80 points or more represents nutritional literacy, and the proportion of patients with nutritional literacy is the level of nutritional literacy. The Cronbach's a coefficient of the scale is 0.893, and the content validity is 0.891, which is considered to be good.
Health-related Quality of Life | Measurements will be conducted before the intervention (baseline measurement), at the end of the intervention (immediate measurement), 3 months after the start of the intervention, and 6 months after the start of the intervention.
  A health-related quality of life scale, the EQ-5D-5L, developed by the EuroQol Group, will be used to measure individuals quality of life. It comprises the EQ-5D descriptive system and the EQ-5D Visual Analog Scale (EQ VAS). The five dimensions assess participants' mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with each dimension having five levels: no difficulties, slight difficulties, moderate difficulties, severe difficulties, and extreme difficulties/unable to perform. the Ul scores ranged from -0.391 to 1. The EQ VAS records a participant's self-assessed health status on a vertical visual analogue scale labelled Your best imagined health (100 points)' and 'Your worst imagined health (0 points)'. The EQ VAS provides a quantitative description of the respondent's perception of their overall health. Higher scores indicate higher quality of life. EQ-5D-5L has been validated by Chinese scholars with a Cronbach coefficient of 0.624.

CONTACTS AND LOCATIONS:
Overall Officials: Meihua Ji, PhD, Principal Investigator — Capital Medical University School of nursing
Locations (4):
- China (4):
  - Songzhuang Community Health Service Center, Beijing, Beijing Municipality
  - Yuqiao Subdistrict Community Health Service Center, Beijing, Beijing Municipality
  - Li Yuan Community Health Service Center in Tongzhou District, Beijing, Beijing, Beijing Municipality
  - Lucheng Subdistrict Community Health Service Center, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weiss BD, Mays MZ, Martz W, Castro KM, DeWalt DA, Pignone MP, Mockbee J, Hale FA. Quick assessment of literacy in primary care: the newest vital sign. Ann Fam Med. 2005 Nov-Dec;3(6):514-22. doi: 10.1370/afm.405. PMID 16338915
- [Result] Luo N, Liu G, Li M, Guan H, Jin X, Rand-Hendriksen K. Estimating an EQ-5D-5L Value Set for China. Value Health. 2017 Apr;20(4):662-669. doi: 10.1016/j.jval.2016.11.016. Epub 2017 Feb 9. PMID 28408009
- [Result] Glasgow RE, Toobert DJ, Barrera M Jr, Strycker LA. The Chronic Illness Resources Survey: cross-validation and sensitivity to intervention. Health Educ Res. 2005 Aug;20(4):402-9. doi: 10.1093/her/cyg140. Epub 2004 Nov 30. PMID 15572438
- [Result] Hill-Briggs F, Gemmell L, Kulkarni B, Klick B, Brancati FL. Associations of patient health-related problem solving with disease control, emergency department visits, and hospitalizations in HIV and diabetes clinic samples. J Gen Intern Med. 2007 May;22(5):649-54. doi: 10.1007/s11606-006-0091-2. PMID 17443373
- [Result] Zhang Y, Zhang Z, Xu M, Aihemaitijiang S, Ye C, Zhu W, Ma G. Development and Validation of a Food and Nutrition Literacy Questionnaire for Chinese Adults. Nutrients. 2022 May 5;14(9):1933. doi: 10.3390/nu14091933. PMID 35565900

DOCUMENTS (1):
  • Informed Consent Form (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT07096102/ICF_001.pdf